CLINICAL TRIAL: NCT00121056
Title: Registry With Enbrel® or Kineret® in a Database Using Longitudinal Evaluations (REKinDLE)
Brief Title: REKinDLE: Registry With Enbrel® or Kineret® in a Database Using Longitudinal Evaluations
Status: Completed | Type: Observational
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Other Study IDs: 20020145
Record Dates: First submitted 2005-06-30; First posted 2005-07-21 (Estimated); Last update posted 2008-12-05 (Estimated); Status verified 2008-12

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etanercept; Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Drug: Enbrel®
Drug: Kineret®

SUMMARY:
The purpose of this study is to determine if Enbrel® or Kineret® will have a positive effect on subject functionality as measured by the Health Assessment Questionnaire Disability Index (HAQDI).

ELIGIBILITY:
Inclusion Criteria: - Subjects with active rheumatoid arthritis as defined by ACR criteria - Able to start Enbrel® or Kineret® therapy (per the approved product monographs) within approximately 30 days of confirmed enrolment Exclusion Criteria: - Active infections at the time of initiating Enbrel® or Kineret® therapy - Malignancy other than basal cell carcinoma of the skin or, in situ carcinoma of the cervix, within the past 5 years - Known hypersensitivity to E. coli derived products - Known hypersensitivity to Enbrel® or any of its components - Subjects receiving, or who received:* Enbrel® in the previous 30 days; * Remicade® in the previous 3 months; * Humira® in the previous 3 months; * Kineret® in the previous 15 days. - Subjects beginning Enbrel® therapy, or treated with prior or current treatment using Enbrel® - Subjects beginning Kineret® therapy, or treated with prior or current treatment using Kineret® - Treatment with any investigational therapy in the 30 days prior to enrolment confirmation - Presence of any significant and uncontrolled medical condition which, in the investigator's opinion, precludes the use of Enbrel® - Sepsis or at risk of septic syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-09

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/08D_FDAMA_113_Posting_Summary_25_IL-1RA_20020145.pdf
- See also: FDA-approved Drug Labeling — http://www.kineretrx.com/